CLINICAL TRIAL: NCT03194984
Title: Randomized Clinical Trial Comparing the Effectiveness of Office Bleaching Agents in Patients of Different Age Group
Brief Title: Effectiveness of Office Bleaching Agents in Patients of Different Age Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Gisele Rodrigues da Silva, professora, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE: 57252216.2.0000.5152
Record Dates: First submitted 2017-05-23; First posted 2017-06-22 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Satisfaction
Keywords: dental whitening; Dental office whitening
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: range of patients aged 18 to 25 years receiving two types of geis and range of patients aged 40-65 years receiving two types of geis
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the patient did not know in which region each gel was applied the investigator did not know in which region each gel was applied the outcomes assessor did not know in which region each gel was applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young Patient (Other): With 18-25 years old. Drug: Hydrogen peroxide 35%. Drug: Hydrogen peroxide 38%
  Interventions: Drug: Hydrogen peroxide 35%; Drug: Hydrogen peroxide 38%
- Adult Patient (Other): With 40-65 years old. Drug: Hydrogen peroxide 35%. Drug: Hydrogen peroxide 38%
  Interventions: Drug: Hydrogen peroxide 35%; Drug: Hydrogen peroxide 38%

INTERVENTIONS:
Drug: Hydrogen peroxide 35% — The office bleaching products will be applied on one of dental hemi-arch of young patients (18-25 years) or adult patients (40-65 years), after randomization. The product will apllied according manufacture instrutions.
  Other Names: Hydrogen peroxide 38%
Drug: Hydrogen peroxide 38% — The office bleaching products will be applied on one of dental hemi-arch of young patients (18-25 years) or adult patients (40-65 years), after randomization. The product will apllied according manufacture instrutions.
  Other Names: Hydrogen peroxide 35%

SUMMARY:
To evaluate the effectiveness in terms of color variation, patient satisfaction, absolute risk and intensity of dentin sensitivity due to dental bleaching in the office with 35% hydrogen peroxide (Whiteness HP Automixx 35%, FGM) and Opalescence Boost 38% ( Ultradent, South Jordan, UT, USA) in the same arch in patients of different age groups: 18 to 25 years and 40 to 65 years. Data will be collected, tabulated and submitted to statistical analysis

DETAILED DESCRIPTION:
Throughout life, the aging of the human being as a whole is inevitable. The dental structure such as cementum and dentin undergo some changes over time, such as secondary deposition of dentin, which results in the reduction of root canal length. In addition, with aging the teeth undergo color changes, presenting a more yellowish or grayish coloration (Ravindra SV et al., 2015). The fact is that most of the studies that involve the technique of dental bleaching have as inclusion factor only young adult patients, excluding patients of more advanced age groups. Therefore, it is fundamental to evaluate the whitening technique in these older patients, since it is a treatment that does not cause harm to the individuals To assess the effect of dental bleaching in the office with Whiteness HP Automixx, FGM at 35% and Opalescence Boost at 38% in the same arch, in different age groups (18 to 25 years and 40 to 65 years) in absolute risk and intensity Of the postoperative dental sensitivity through the visual analog (VAS 0-10) and analogue (NRS 0-4) scales.

* Evaluate the efficacy of Whitening HP Automixx, FGM 35% and Opalescence Boost 38% in the same arch in different age groups (18 to 25 years and 40 to 65 years) using Color Vita Classical and Vita Bleachedguide, and the Vita Easyshade spectrophotometer.
* Evaluate the satisfaction of patients after Whitening HP Automixx at 35, FGM and Opalescence Boost 38% in the same arch in different age groups (18 to 25 years and 40 to 65 years).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age up to 25 years
* Patients aged 40 years up to 65 years
* Good oral and general health
* Teeth free of restorations or with small restorations
* Free from carious injury,
* Patients with tooth color A2 or darker according to the Vita Classical color scale (Vita Zahnfabrik, Bad Säckingen, Germany)
* Agree to the informed consent form

Exclusion Criteria:

* extensive restoration
* Patients who have already undergone dental whitening
* Pregnant or lactating women
* That report dental sensitivity
* With non-carious cervical lesion
* Parafunctional habits
* Orthodontic appliances
* Any other type of oral pathology
* Smokers, patients who are using analgesic or anti-inflammatory drugs, present systemic alterations such as gastric, cardiac, renal and hepatic problems, diabetics, hypertensives or pre-existing neoplasias.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Tooth discoloration | 36 weeks
  Efficacy of office dental whitening mensured by Easyshade spectrophotometer.

SECONDARY OUTCOMES:
Dentin sensitivity | 36 weeks
  It will analised the risk and intensity of tooth sensitivity of dental bleaching
Patient satisfaction | 36 weeks
  It will analised the patient satisfaction by questionnaire of self-perception of aesthetics (PIDAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Gisele Silva, Dra, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Gisele Rodrigues da Silva, Uberlândia, Av Pará S/n Bloco 4 L Anexo A Sala 42 Campus Umuarama, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Geus JL, Wambier LM, Kossatz S, Loguercio AD, Reis A. At-home vs In-office Bleaching: A Systematic Review and Meta-analysis. Oper Dent. 2016 Jul-Aug;41(4):341-56. doi: 10.2341/15-287-LIT. Epub 2016 Apr 5. PMID 27045285
- [Background] Kossatz S, Dalanhol AP, Cunha T, Loguercio A, Reis A. Effect of light activation on tooth sensitivity after in-office bleaching. Oper Dent. 2011 May-Jun;36(3):251-7. doi: 10.2341/10-289-C. Epub 2011 Jul 8. PMID 21740236
- [Background] Reis A, Dalanhol AP, Cunha TS, Kossatz S, Loguercio AD. Assessment of tooth sensitivity using a desensitizer before light-activated bleaching. Oper Dent. 2011 Jan-Feb;36(1):12-7. doi: 10.2341/10-148-CR. Epub 2011 Mar 24. PMID 21488723
- [Background] Martin J, Rivas V, Vildosola P, Moncada L, Oliveira Junior OB, Saad JR, Fernandez E, Moncada G. Personality Style in Patients Looking for Tooth Bleaching and Its Correlation with Treatment Satisfaction. Braz Dent J. 2016 Jan-Feb;27(1):60-5. doi: 10.1590/0103-6440201600127. PMID 27007348
- Available data/document: Metanalysis, systematic review: 27045285 — https://www.ncbi.nlm.nih.gov/pubmed/?term=27045285
- Available data/document: Clinical Study Report: 21740236 — https://www.ncbi.nlm.nih.gov/pubmed/?term=21740236
- Available data/document: Clinical Study Report: 21488723 — https://www.ncbi.nlm.nih.gov/pubmed/?term=21488723
- Available data/document: Informed Consent Form: 27007348 — https://www.ncbi.nlm.nih.gov/pubmed/?term=27007348